CLINICAL TRIAL: NCT00226395
Title: Randomized, Double-Blind, Placebo- and Active-Control, Single- and Multiple-Dose Evaluation of the Analgesic Efficacy and Safety of Oxymorphone Immediate Release (IR) Tablets in Patients With Moderate/Severe Pain Following Abdominal Surgery
Brief Title: Efficacy and Safety of Oxymorphone Immediate Release in Post-surgical Acute Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3203-009
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Acute Pain
Keywords: oxymorphone; acute pain; abdominal surgery; opioids
MeSH Terms: conditions — Acute Pain | interventions — Oxymorphone

INTERVENTIONS:
Drug: Oxymorphone immediate release

SUMMARY:
The purpose of this study is to evaluate the analgesic efficacy and safety of two doses of oxymorphone immediate release (IR) compared to placebo and oxycodone in post-surgical pain.

DETAILED DESCRIPTION:
Following abdominal surgery and after sufficient washout from post-surgical analgesia, patients were randomized to one of the following four treatment groups; 1) oxymorphone IR 10 mg, 2) oxymorphone IR 20 mg, 3) oxycodone IR 15 mg, or 4) placebo. Total duration of treatment was 48 hours. Patients were required to take the study medication every 4-6 hours. After the first dose, periodic pain assessments were performed for the first six hours. Subsequently, patients were required to assess their current pain intensity and average pain intensity since the last dose of study medication just prior to every dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older
* Patients undergoing surgery through an abdominal incision of at least 3 cm who are expected to be hospitalized for at least 36 hours and are expected to subsequently require at least 48 hours of oral opioid therapy.
* Washout of at least 45 minutes for parenteral and 4 hours for IM analgesia.
* Initial pain intensity score of at least 50 mm on a 100-mm VAS and a categorical pain rating of moderate or severe on a scale of none, mild, moderate, or severe.
* Written informed consent.

Exclusion Criteria:

* Known allergy or significant reaction to opioids.
* History of chronic opioid use or opioid abuse within 6 months prior to study entry.
* History of alcohol or substance abuse within the last 3 years.
* Have been a participant in a study of an investigational drug or device within 30 days prior to study entry.
* Have been a previous participant in an oxymorphone clinical trial.
* Are currently taking or have taken a monoamine oxidase inhibitor (MAOI) drug within 2 weeks prior to study entry.
* Are currently taking or have taken St. John's Wort >1000 mg/day within 2 days prior to study entry.
* Use of long-acting oral and parenteral analgesics (opioid, non-opioid or non-steroidal anti-inflammatory drug [NSAID]) within 12 hours (at least 24 hours for cyclooxygenase-2 [COX 2] analgesics) prior to receiving study medication.
* Are not stabilized on the following medications for at least 4 weeks prior to dosing: tricyclic antidepressant drugs; serotonin reuptake inhibitors; amphetamines used for attention-deficit hyperactivity disorder (ADHD)
* Have a history of seizure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2004-09; Study Completion 2005-08

PRIMARY OUTCOMES:
Time to discontinuation due to all causes

SECONDARY OUTCOMES:
The following are the secondary endpoints during the initial 6 hours following the first dose of study medication:
- 6-Hour Sum of Pain Intensity Differences (SPID; VAS and categorical)
- 6-Hour Total Pain Relief Scores (TOTPAR; VAS and categorical)
- Time (in hours) to First Perceptible Pain Relief
- Time (in hours) to Meaningful Pain Relief
- Hourly Pain Relief Scores
- Hourly Pain Intensity Difference Scores
The following are the secondary endpoints during the multiple dosing phase:
- Mean average pain intensity scores collected during the dosing intervals.
- Mean current pain intensity (VAS) collected during the dosing intervals.
- Patient's global evaluation of study medication at the end of study.
- Physician's global evaluation of study medication at the end of study.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Brookwood Medical Center, Birmingham, Alabama
  - The Medical Center, Dept. Clinical research, Birmingham, Alabama
  - Montgomery Women's Health Associates, Montgomery, Alabama
  - Arrowhead Community Hospital, Phoenix, Arizona
  - John C Lincoln Hospital, Phoenix, Arizona
  - Paradise Valley Hospital, Phoenix, Arizona
  - Glendale Adventist Medical Center, Glendale, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Huntington Memorial Hospital, Pasadena, California
  - Palm West Hospital, Palm Springs, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Medical Park Hospital, Winston-Salem, North Carolina
  - Univ. Pittsburgh Hospital, Pittsburgh, Pennsylvania
  - Univ. Pittsburgh Medical center, Pittsburgh, Pennsylvania
  - Memorial Hermann Memorial City Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Cottonwood Hospital, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - McKay-Dee Hospital, Salt Lake City, Utah